CLINICAL TRIAL: NCT03768193
Title: Comparison of Ultrasound-guided Continuous Serratus Anterior Plane Blockade With Continuous Thoracic Paravertebral Blockade for Perioperative Analgesia Following Video-assisted Thoracoscopic Surgery (VATS)
Brief Title: Deep Serratus Anterior Plane Block vs Surgically-placed Paravertebral Block for VATS Surgery
Acronym: SAPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Dr Conor Hearty, Consultant Anaesthetist, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/378/1918
Record Dates: First submitted 2018-09-27; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Thoracic Diseases; Thoracic Surgery; Rib Fractures; Pain, Postoperative; Pain, Procedural; Anaesthesia, Regional
MeSH Terms: conditions — Thoracic Diseases; Rib Fractures; Pain, Postoperative; Pain, Procedural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep serratus anterior plane block (Experimental): Ultrasound-guided deposition of 40mls of 2mg/ kg levobupivacaine into the deep serratus anterior plane space, in the mid axillary line, at the level of the 4th/5th rib. Insertion of a continuous local anaesthetic infusion catheter(Portex™) and continuation of an infusion of 0.125% levobupivacaine at a rate of 8-12mls/ hour for 48 hours.
  Interventions: Procedure: Deep serratus anterior plane block
- Surgically-placed paravertebral block (Active Comparator): Surgical placement of paravertebral local anaesthetic infusion catheters (Portex™) prior to closure. Bolus of levobupivacaine as per protocol. Continuation of an infusion of 0.125% levobupivacaine at a rate of 8-12mls/ hour for 48 hours.
  Interventions: Procedure: Surgically-placed paravertebral block

INTERVENTIONS:
Procedure: Deep serratus anterior plane block — Deposition of local anaesthetic in the space between the serratus anterior muscle and the external intercostal muscle, at the level of the 4th-5th rib, in the midaxillary line. Procedure performed under ultrasound guidance. Catheter - based infusion of local anaesthetic into this space for 48 hours.
  Arms: Deep serratus anterior plane block
Procedure: Surgically-placed paravertebral block — Surgically-placed paravertebral block catheters for continuous local anaesthetic infusion of 0.125% levobupivacaine at 8-12mls/ hr for 48 hours.
  Arms: Surgically-placed paravertebral block

SUMMARY:
Thoracic surgery, and surgery involving the chest wall in general, is associated with poorly controlled acute pain, which may result in delayed functional recovery, and may progress to chronic pain. Multimodal opioid-sparing analgesia regimens are a key component of the thoracic surgery enhanced recovery pathway, the aim of which is to improve outcomes in patients undergoing both minimally invasive and open thoracic surgical procedures. Novel interfascial plane blocks are emerging as feasible alternatives to central neuraxial analgesia techniques in a variety of clinical settings.

The aim of this study is to show non-inferiority of serratus anterior blockade compared with surgically placed paravertebral blocks in the management of perioperative acute pain in patients undergoing VATS procedures.

DETAILED DESCRIPTION:
Post-thoracotomy pain syndrome is an unwanted complication of thoracic surgery. Poorly controlled pain may precipitate increased morbidity in the immediate and early postoperative periods due to its adverse effects on respiratory mechanics and mobilisation, which may result in further morbidity such as postoperative pulmonary complications and thrombosis. Poor perioperative management of this pain may also result in the development of chronic pain. Enhanced recovery, particularly functional recovery has become an important goal in the perioperative management of our patients. A key principle of this pathway is multimodal opioid-sparing analgesia to facilitate improved recovery and patient outcomes. Regional anaesthesia forms the cornerstone of this multimodal analgesia regimen.

Traditionally, thoracic epidural and thoracic paravertebral blockade have been the main forms of regional anaesthesia utilised in thoracic surgical patients undergoing lung resection. With the increasing use of minimally invasive thoracic surgery and with a cohort of patients who may not always be suitable for central neuraxial blockade, alternatives are needed. More recently, there has been an emerging use of interfascial plane blocks in this patient group. The interest in these techniques is derived from case reports, case series, cadaveric studies, and small clinical trials, which have demonstrated clinical efficacy in a variety of elective and emergency thoracic surgical procedures and also in chronic thoracic pain syndromes.

The deep serratus anterior plane (deep SAP) block is a relatively new interfascial plane regional anaesthesia technique, which has been postulated to provide analgesia of the entire hemithorax. The mechanism of its analgesic effects are believed to occur via blockade of the lateral cutaneous branches of the thoracic intercostal nerves (T2-T12), which produces analgesia of the anterolateral chest wall. A recent anatomical study by Mayes et al. demonstrated consistent blockade of the lateral cutaneous branches of the intercostal nerves. Clinical studies, although small, have shown dermatomal spread in the T2 - T9 distribution of the anterolateral chest wall. Therefore, this block presents a potential alternative to central neuraxial blockade.

However, whether SAP blockade can produce non-inferior analgesia compared with either thoracic epidural or thoracic paravertebral, both in terms of somatic +/- autonomic blockade, and the reliability of dermatomal spread, has been questioned by some.

The aim of this randomised controlled trial is to demonstrate non-inferiority of ultrasound-guided continuous deep serratus anterior plane blockade compared with surgically-placed continuous paravertebral blockade, for perioperative analgesia, in the patients undergoing minimally-invasive videoscopic thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

• All adults greater than or equal to 18 years of age presenting for minimally-invasive thoracic surgery.

Exclusion Criteria:

* Patient refusal.
* Local infection at site of insertion.
* Allergy to amide local anaesthetics, opioids, paracetamol, NSAIDs, ketamine, NMBs, volatile anaesthetics.
* Concurrent use of antiarrhythmics with local anaesthetic activity.
* Concurrent use of MAOIs or within 2 weeks of MAOI use.
* Severe renal, liver or cardiac dysfunction.
* Coagulopathy/ anticoagulants that preclude use of PVB/ SAP techniques.
* Inability to comprehend pain scoring system.
* Elderly or frail patients that require a reduction in levobupivacaine dose commensurate with their physical status, resulting in the protocol not being followed.
* Pregnancy, breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Over the first 48 hours postoperatively
  Expressed as oral morphine equivalent

SECONDARY OUTCOMES:
Postoperative numerical pain scores | Over the first 48 hours postoperatively
  Numerical rating scale. 0 - 10. 0=no pain, 1-3=mild pain, 4-6=moderate pain, 7-10=severe pain.
Opioid side - effects - 1 | Over the first 48 hours postoperatively
  Sedation scale. 0 = wide awake, 1 = drowsy but responds to normal verbal communication, 2 = asleep, but awakes with verbal communication. 3 = asleep, awakens with mild physical stimulation. 4 = asleep, unresponsive to physical stimulation.
Opioid side - effects - 2 | Over the first 48 hours postoperatively
  Nausea/ vomiting scale. Questionnaire. 0= none, 1=mild, 2=moderate, 3=severe
Opioid side - effects - 3 | Over the first 48 hours postoperatively
  Itch/ Pruritis scale 0= none, 1=mild, 2=moderate, 3=severe
Mean arterial blood pressure | Over the first 48 hours postoperatively.
  Calculated from systolic and diastolic blood pressure.
Presence of dermatomal sensory block distribution | Within the first 24 hours postoperatively
  Dermatomal sensory block distribution
Functional assessment | Within the first 48 hours postoperatively
  Walking distance in meters assessed by physiotherapist
Patient satisfaction | Over the first 48 hours postoperatively
  Subjective patient satisfaction scale. Subjective scale assessing Level of overall patient satisfaction with perioperative analgesia. Patient rates their experience as either 1 = insufficient, 2 = sufficient, 3 = very good, 4 =excellent.
Duration of inpatient hospital admission | From date of admission for surgery to date of discharge by the thoracic team; through to study completion.
  Measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Hearty, FFPMCAI,FFPMANZCA,FCARCSI,FIPP, Principal Investigator — Consultant Anaesthetist, Mater Misericordiae University Hospital
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Hanley C, Wall T, Bukowska I, Redmond K, Eaton D, Ni Mhuircheartaigh R, Hearty C. Ultrasound-guided continuous deep serratus anterior plane block versus continuous thoracic paravertebral block for perioperative analgesia in videoscopic-assisted thoracic surgery. Eur J Pain. 2020 Apr;24(4):828-838. doi: 10.1002/ejp.1533. Epub 2020 Jan 30. PMID 31955478